CLINICAL TRIAL: NCT06346145
Title: A Randomized Controlled Trial Comparing Metabolic Surgery to Standard Care in Patients With Severe Obesity and Established Cardiovascular Disease
Brief Title: Impact of Bariatric Surgery on Heart Disease Compared to Standard Care
Acronym: MIMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danderyd Hospital (Other)
Collaborators: Karolinska Institutet (Other); The 21 healthcare regions in Sweden (Unknown)
Responsible Party: Principal Investigator, Erik Näslund, Professor, Danderyd Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIMS study; 2023-00453 (Other Grant/Funding Number: Swdeish research council)
Record Dates: First submitted 2024-03-15; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Obesity, Morbid; Bariatric Surgery Candidate; Heart Diseases
MeSH Terms: conditions — Obesity, Morbid; Heart Diseases | interventions — Bariatric Surgery; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bariatric surgery (Active Comparator): Gastric bypass or gastric sleeve
  Interventions: Procedure: Bariatric surgery
- Standard care (Active Comparator): Standard obesity treatment offered in Swedish regions
  Interventions: Procedure: Standard care

INTERVENTIONS:
Procedure: Bariatric surgery — Type of surgery assigned by surgeon in consultation with patient
  Arms: Bariatric surgery
Procedure: Standard care — Standard care can consist of dietary intervention, physiotherapy or drug treatment in accordance to the care given in the region of Sweden where the patient resides.
  Arms: Standard care

SUMMARY:
Obesity is associated with type 2 diabetes (T2D) and cardiovascular disease (CVD). Metabolic and bariatric surgery (MBS) has in several randomized controlled trials (RCT) been shown to be superior to best medical therapy in the treatment of T2D. In the area of CVD, RCT after MBS are lacking. It was recently demonstrated in a cohort study that MBS in patients with severe obesity and a previous myocardial infarction (MI) was associated with a 50% reduction in the risk of death and new MI. The aim of this proposal is to confirm this in a nationwide RCT. Using the nationwide SWEDEHEART database patients with severe obesity and a previous MI will be identified. They will be contacted and offered participation. After informed consent the patients will be randomized to MBS or optimized care (including visit with a cardiologist and optimization of secondary preventive measures and referral to dietician/physiotherapist). The primary outcome measure is a major cardiovascular adverse event (MACE). Secondary outcome measures include mortality, new MI, stroke, heart failure and atrial fibrillation. Tertiary outcome measures include health related quality of life and surgical complications. Patients will be followed in the nationwide metabolic surgery register SOReg, the national inpatient register, national cause of death register, the Swedish prescribed drug register, and the Swedish population register. If positive results these can be included in guidelines for MBS.

ELIGIBILITY:
Inclusion Criteria:

* MI (as defined by the universal definition of MI) at least 1 year before inclusion.
* BMI ≥35 kg/m2
* Written informed consent obtained

Exclusion Criteria:

* Any condition that may influence the patient's ability to comply with study protocol.
* Earlier MBS or operation for gastric or duodenal ulcer or reflux disease
* Other condition that makes patient not suitable for MBS according to responsible surgeon and anesthesiologist
* Unable to understand Swedish.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
MACE defined as first occurrence of death (all-cause mortality), MI, stroke, myocardial revascularization (not related to MI), hospital admission because of heart failure or atrial fibrillation as a primary ICD diagnosis. | Through study completion, expected average of 6 years
  Data will be obtained for the Swedish national patient registry and other national quality registries.

SECONDARY OUTCOMES:
Total event rate | Through study completion, expected average of 6 years
  Based on events listed in the primary outcome measure. Data will be obtained for the Swedish national patient registry and other national quality registries.
All-cause mortality | Through study completion, expected average of 6 years
  Data will be obtained for the Swedish national national quality registries.
Cardiovascular death | Through study completion, expected average of 6 years
  Data will be obtained for the Swedish national national quality registries.
Remission of type 2 diabetes (T2D) and hypertension | Through study completion, expected average of 6 years
  Number of patients in remission
Myocardial infarction | Through study completion, expected average of 6 years
  Data will be obtained for the Swedish national national quality registries.
Stroke | Through study completion, expected average of 6 years
  Data will be obtained for the Swedish national national quality registries.
Myocardial revascularization (not related to MI) | Through study completion, expected average of 6 years
  Data will be obtained for the Swedish national national quality registries.
hospital admission because of heart failure as a primary ICD diagnosis. | Through study completion, expected average of 6 years
  Data will be obtained for the Swedish national national quality registries.
hospital admission because of atrial fibrillation as a primary ICD diagnosis. | Through study completion, expected average of 6 years
  Data will be obtained for the Swedish national national quality registries.

OTHER OUTCOMES:
Safety, i.e., no excess of severe complications (Clavien-Dindo ≥3b (a complication requiring intervention under general anesthesia or resulting in organ failure or death)) and long-term morbidity. | Through study completion, expected average of 6 years
  Data will be obtained for the Swedish national patient registry and other national quality registries.
Body weight change | 5-year follow-up
  Change in kg from baseline during long-term follow-up.
Change in quality of life | 5-year follow-up
  Assessed by EQ-5D-5L questionnaire
All-cause hospitalizations | Through study completion, expected average of 6 years
  Based on ICD 10 diagnosis in national patient registry and other national quality registries
Change in quality of life | 5-year follow-up
  Assessed by RAND 36

CONTACTS AND LOCATIONS:
Overall Officials: Erik Näslund, MD, PhD, Principal Investigator — Karolinska Institutet/Danderyd hospital

IPD SHARING:
Plan to Share IPD: No
Data will not be shared openly at a repository since it contains personal data. Data will be made available upon request after ensuring compliance with relevant legislation and Karolinska Institutet guidelines.

REFERENCES:
- [Background] Naslund E, Stenberg E, Hofmann R, Ottosson J, Sundbom M, Marsk R, Svensson P, Szummer K, Jernberg T. Association of Metabolic Surgery With Major Adverse Cardiovascular Outcomes in Patients With Previous Myocardial Infarction and Severe Obesity: A Nationwide Cohort Study. Circulation. 2021 Apr 13;143(15):1458-1467. doi: 10.1161/CIRCULATIONAHA.120.048585. Epub 2020 Oct 26. PMID 33103469